CLINICAL TRIAL: NCT03609606
Title: An Open-label, Randomized, Multiple-dose Crossover Study to Investigate Drug Interaction Between D326, D337, and D013 in Healthy Male Subjects
Brief Title: A Study to Investigate Drug Interaction Between D326, D337, and D013 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 183DDI18011
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Dyslipidemias; Hypertension
Keywords: Dyslipidemia; Hypertension; CKD-386; Drug-Drug Interaction
MeSH Terms: conditions — Dyslipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A, Sequence1 (Experimental): * Period 1: Treatment of D013, D326 and D337 on Day1~Day7
  * Period 2: Treatment of D013 on Day22~Day28
  Interventions: Drug: D013, D326 and D337; Drug: D013
- Part A, Sequence 2 (Experimental): * Period 1: Treatment of D013 on Day1~Day7
  * Period 2: Treatment of D013, D326 and D337 on Day22~Day28
  Interventions: Drug: D013, D326 and D337; Drug: D013
- Part B, Sequence 1 (Experimental): * Period 1: Treatment of D013, D326 and D337 on Day1~Day7
  * Period 2: Treatment of D326 and D337 on Day22~Day28
  Interventions: Drug: D013, D326 and D337; Drug: D326 and D337
- Part B, Sequence 2 (Experimental): * Period 1: Treatment of D326 and D337 on Day1~Day7
  * Period 2: Treatment of D013, D326 and D337 on Day22~Day28
  Interventions: Drug: D013, D326 and D337; Drug: D326 and D337

INTERVENTIONS:
Drug: D013, D326 and D337 — Daily oral administration of 1 tablet for each drug under fasting conditions for 7 days
  Other Names: CKD-386 Test
Drug: D013 — Daily oral administration of 1 tablet under fasting conditions for 7 days
  Other Names: CKD-386 Reference1
  Arms: Part A, Sequence 2; Part A, Sequence1
Drug: D326 and D337 — Daily oral administration of 1 tablet for each drug under fasting conditions for 7 days
  Other Names: CKD-386 Reference2
  Arms: Part B, Sequence 1; Part B, Sequence 2

SUMMARY:
A study to investigate drug interaction between D326, D337, and D013 in healthy male subjects

DETAILED DESCRIPTION:
An open-label, randomized, multiple-dose crossover study to investigate drug interaction between D326, D337, and D013 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between ≥ 20 and ≤ 45 years old
2. Weight ≥ 50kg, with calculated body mass index(BMI) of ≥ 18 and ≤ 29.9kg/m²
3. Subjects who agree to use a combination of effective contraceptive methods or medically acceptable contraceptive methods for up to 28 days after the date of administration of the clinical trial drug and agree not to provide sperm
4. Subject who are informed of the investigational nature of this study, voluntarily agree to participate in this study

Exclusion Criteria:

1. History or presence of clinically significant and active cardiovascular, respiratory, hepatobiliary, renal, hematological, gastrointestinal, endocrine, immune, dermatologic, neurologic or psychiatric disorder
2. With symptoms indicating acute illness within 28 days prior to the first Investigational Product administration
3. Any medical history that may affect drug absorption, distribution, metabolism and excretion
4. Genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose uptake disorder
5. Any clinically significant active chronic disease

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
AUCtau(area under the plasma concentration-time curve for a dosing interval at steady state) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing
Cmax,ss(Maximum plasma concentration of the drug at steady state) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing

SECONDARY OUTCOMES:
Cmin,ss(Minimum concentration of the drug in plasma at steady state) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing
Tmax,ss(Time to maximum plasma concentration at steady state) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing
t1/2(Terminal elimination half-life) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing
CLss/F(Apparent total body clearance of the drug from plasma at steady state) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing
Vd,ss/F(Apparent volume of distribution at steady state) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing
PTF(Peak-to-trough fluctuation) | 0(predose)~24 hours at Day7 and Day28
  * Part A: Pharmacokinetic parameter of D013 after multiple dosing
  * Part B: Pharmacokinetic parameters of D326 and D337 after multiple dosing

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, M.D., Ph.D, Principal Investigator — Department of Pharmacology, College of Medicine/ Department of Clinical Pharmacology&Toxicology, Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No